CLINICAL TRIAL: NCT00786097
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability, Dermical Sensitivity) of Dermacyd PH_DETINLYN (Lactic Acid) Tangerine Mix
Brief Title: Dermacyd PH_DETINLYN (Lactic Acid) Tangerine Mix - Compatibility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04305
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Dermacyd PH_DETINLYN (Lactic Acid)
  Interventions: Drug: Dermacyd PH_DETINLYN (Lactic Acid)

INTERVENTIONS:
Drug: Dermacyd PH_DETINLYN (Lactic Acid)

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd PHDETINLYN Tangerine Mix.None.

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin I,II, III e IV
* Integral skin test in the region;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion inclusion:

* Lactation or gestation
* Use of Antiinflammatory and/or immunossupression drugs
* Personnel history of atopy;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease;
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermical irritability and dermical sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil